CLINICAL TRIAL: NCT06073470
Title: Exploration of the Metabolic Mechanisms of the Electrophysiological Biomarkers for Response to Methylphenidate Treatment in Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: Metabolic Mechanisms of the Electrophysiological Biomarkers for Response to Methylphenidate Treatment in Children With ADHD
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202204054RINC
Record Dates: First submitted 2023-09-15; First posted 2023-10-10 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-09

CONDITIONS: Methylphenidate; Metabolomics
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD GROUP: Subjects with clinical diagnosis of ADHD according to the DSM-V criteria
  Interventions: Drug: methylphenidate
- TD GROUP: Typically development controls without lifetime diagnosis with ADHD

INTERVENTIONS:
Drug: methylphenidate — The patients with ADHD will receive 12-week treatment with methylphenidate.
  Groups: ADHD GROUP

SUMMARY:
To explore the relationship of treatment-related changes in electrophysiology and those in metabolomics for identification of the underlying metabolic mechanisms for the electrophysiological effects of methylphenidate in children with ADHD.

DETAILED DESCRIPTION:
Although the efficacy of methylphenidate in reducing the core symptoms of attentiondeficit/ hyperactivity disorder (ADHD) is well documented in clinical trials, no definite biomarker has been identified to differentiate responders from non-responders to methylphenidate treatment for children with ADHD. In addition, the neural and metabolic mechanisms underlying the therapeutic effects of methylphenidate remain to be elucidated. In this 4-year prospective project, the investigators will explore the effects of 12-week treatment with methylphenidate on the electrophysiology and metabolomics of children with ADHD to identify the biomarkers for predicting the clinical response to methylphenidate. In addition, the investigators will explore the metabolic mechanisms through which methylphenidate treatment may modulate the abnormality in the electrophysiology of children with ADHD.

Specific Aims:

1. To examine the differences in electrophysiology and metabolomics between children with ADHD and neurotypical controls.
2. To examine the differences in the change of electrophysiology and metabolomics after 12-week treatment with methylphenidate between responders and non-responders in children with ADHD.
3. To explore the relationship of treatment-related changes in electrophysiology and those in metabolomics for identification of the underlying metabolic mechanisms for the electrophysiological effects of methylphenidate in children with ADHD.

ELIGIBILITY:
1. Patients with ADHD

   1. Inclusion Criteria

      * Patients, aged 6 to 18 years, meet the DSM-5 diagnostic criteria for ADHD.
      * At baseline, patients have a Clinical Global Impressions-ADHD-Severity (CGI-ADHD-S) score greater than 4.
      * Patients have a Full IQ (FIQ) score greater than 80.
   2. Exclusion Criteria

      * Patients have a major psychiatric disorder, such as autism spectrum disorder, schizophrenia, affective disorders, or substance use disorders.
      * Patients have a major disorder of central nervous system, such as epilepsy.
      * Patients have a major systemic disease, such as diabetes mellitus or cardiovascular diseases.
      * Patients have ever received any medication to treat the clinical symptoms of ADHD.
2. Neurotypical participants:

   1. Inclusion Criteria

      * aged 6 to 18 years
      * All of the neurotypical participants have no psychiatric disorder in lifetime according to the diagnostic criteria of DSM-5.
   2. Exclusion Criteria

      * participants have any disorder of central nervous system or major systemic disease
      * participants have ever taken any psychotropic drug, or who have FIQ scores less than 80, will be excluded from the present study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 80drug-naïve patients with ADHD, aged 6-18, and 80 age- and sex-matched typically developing controls will be recruited in this project
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic interview | 1 hour
  We will interview all the participants and their parents to examine whether the participants have any psychiatric disorder by employing the Kiddie Epidemiologic version of the Schedule for Affective Disorders and Schizophrenia (K-SADS-E).
ADHD symptoms | 15 minutes
  Subjects will be interviewed by ADHD rating scale , which consists of 18 items to measure the symptomatology of ADHD . Each question in this questionnaire is scaled from 0 to 3. The higher the total score, the more severe the symptoms.

SECONDARY OUTCOMES:
Questionnaire | 5minutes
  Cases and parents assisted in filling out the Achenbach child behavior check list (CBCL).Each question in this questionnaire is scaled from 1 to 3. The higher the total score, the more severe the emotional and behavioral distress.
Questionnaire | 5minutes
  Cases and parents assisted in filling out the Swanson, Nolan, and Pelham Rating Scale Fourth Edition (SNAP-IV).Each question in this questionnaire is scaled from 0 to 3. The higher the total score, the more severe the symptoms.
Questionnaire | 5minutes
  Cases and parents assisted in filling out the Family APGAR questionnaire.Each question in this questionnaire is scaled from 0 to 2. The higher the total score, the better the family function.
Questionnaire | 5minutes
  Cases and parents assisted in filling out the Social Adjustment Inventory for Children and Adolescents questionnaire (SAICA).The scale for each question in this questionnaire ranges from 1 to 4. The higher the total score, the worse the social adaptation status.
Questionnaire | 5minutes
  Cases and parents assisted in filling out the Behavior Rating Inventory of Executive Function questionnaire(BRIEF).Each question in this questionnaire is scaled from 1 to 3. The higher the total score, the lower the executive function status.
Neurobiological assessments | 10minutes
  Resting state EEG will be recorded in NTUH ERP lab.The EEG will be processed for functional connectivity indices between regions are calculated using the magnitude squared coherence (Coh) in the delta(delta)/theta(theta)/alpha(alpha)/beta(beta) frequency bands and the nonlinear index (L) of generalized synchronization.
Neurobiological assessments | 10minutes
  Resting state EEG will be recorded in NTUH ERP lab. Phase transfer entropy (PTE) will be used to construct the effective connectivity. The topological properties of networks and flow gain are measured separately in four bands (delta, theta, alpha, and beta).
Neurobiological assessments | 10minutes
  Resting state EEG will be recorded in NTUH ERP lab. We will perform Fast Fourier Transform using the pwelch algorithm, with a 128 sample triangular window, to obtain time-frequency domain measures. Mean spectral estimates in various power bands are computed. As a measure of intraindividual variability in neural activity, the standard deviation of the power in each 2-second trial is calculated for each band for each participant.
Neurobiological assessments | 30minutes
  auditory MMN/P3a (task-free ERP) will be recorded in NTUH ERP .
Neurobiological assessments | 20minutes
  dichotic continuous performance task(DCPT, task-related ERP modified from Conner's CATA) will be recorded in NTUH ERP lab.
liquid chromatography-mass spectrometry and gas chromatography-mass spectrometry | 5 minutes
  Whole blood samples will be collected after 8 hours of fasting at baseline and week 12 for neurotypical controls and for patients with ADHD. The investigators will employ both liquid chromatography coupled to mass spectrometry (LC/MS) and gas chromatography coupled to mass spectrometry (GC/MS) to conduct the experiments of metabolomic profiling of the serum at the Metabolomics Core Laboratory, National Taiwan University.
Neuropsychological testing | 1.5 hours
  Subjects will be assessed by the WISC-V(Wechsler Intelligence Scale for Children),WISC-V scores between 90 and 109 represent moderate general intelligence, and higher scores represent relatively better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Study Director — Department of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan